CLINICAL TRIAL: NCT00994110
Title: Prospective Randomized, Double Blind, Placebo Controlled Trial of SOM230 for the Reduction of Post-Pancreatectomy Fistula, Leak, and Abscess
Brief Title: Placebo Controlled Trial of SOM230 for the Reduction of Post-Pancreatectomy Fistula, Leak, and Abscess
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-039
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Pancreatic Cancer
Keywords: PANCREAS; Pasireotide; SOM230; saline placebo; 09-039
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- SOM230 (Experimental): This is a randomized, double-blind, placebo controlled phase III trial of SOM230 vs. saline placebo in patients undergoing pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy at Memorial Sloan-Kettering Cancer Center.
  Interventions: Drug: Pasireotide (SOM230)
- placebo (Placebo Comparator): This is a randomized, double-blind, placebo controlled phase III trial of SOM230 vs. saline placebo in patients undergoing pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy at Memorial Sloan-Kettering Cancer Center.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Pasireotide (SOM230) — Patients will receive subcutaneous injection of SOM230 or placebo (NS, equivalent volume) on the day of operation prior to resection in the pre-surgical center. The initial subcutaneous injection of drug or placebo will be given at least one hour prior but no longer than 8 hours prior to transection of the pancreas. Patients will be continuously monitored in the OR following this dose administration, and both their cardiac and respiratory status will be closely followed.
  Postoperatively patients will receive study drug or placebo every 12 hours. Subcutaneous injections will continue until postoperative day 7, with the last dose administered in the evening on postoperative day 6, or until a pancreatic complication has been identified.
  Arms: SOM230
Other: placebo — Patients will receive subcutaneous injection of SOM230 or placebo (NS, equivalent volume) on the day of operation prior to resection in the pre-surgical center. The initial subcutaneous injection of drug or placebo will be given at least one hour prior but no longer than 8 hours prior to transection of the pancreas. Patients will be continuously monitored in the OR following this dose administration, and both their cardiac and respiratory status will be closely followed.
  Postoperatively patients will receive study drug or placebo every 12 hours. Subcutaneous injections will continue until postoperative day 7, with the last dose administered in the evening on postoperative day 6, or until a pancreatic complication has been identified.
  Arms: placebo

SUMMARY:
The purpose of this study is to help us learn more about how to lower the patient's risk of the most common complications after their pancreas operation. After tumors are removed and the remaining part of the pancreas is connected to the intestine or closed, a leakage of pancreatic fluid may occur. This fluid may form an "abscess" (collection of pus) or "fistula" that would need to be drained. A fistula is a persistent leakage of pancreatic fluid that sometimes occurs after pancreatic surgery. Fistulas, leaks, and abscesses are complications that are seen in roughly every 15-20 patients out of every 100 that have pancreas surgeries. Complications like these extend the patient's stay in the hospital after surgery. These complications may require the patient's doctor to perform additional tests or procedures to treat them.

The physical and emotional burden these complications place upon patients, as well as the financial cost to the health care system, can be great. The surgeons at Memorial Sloan-Kettering Cancer Center are conducting a study to determine if a drug, SOM230, can help reduce the rate of these complications. SOM230, also known as Pasireotide, is a drug that has been observed to reduce the rate of similar complications in other studies.

The surgeon would like to compare the effects, good and/or bad, of SOM230 with "placebo" (solution without medication) to see if SOM230 reduces the rate of fistulas, leaks and abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or greater.
* Signed informed consent
* Candidate for pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy.

Exclusion Criteria:

* Pregnancy
* Patients with malabsorption syndrome, short bowel or chologenic diarrhea not controlled by specific therapeutic means.
* Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 250mg/dl.

Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.

* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment.
* Patients who are at risk for QT prolongation. Risk factors include: patients with electrolyte disturbances such as hypokalemia, hypomagnesemia, and hypocalcemia; patients with a family history of long QT syndrome. syncope, and idiopathic sudden death; patients with concomitant diseases that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism, bradycardia, high-grade AV block, significant cardiac arrhythmias, or cardiac failure; patients using concomitant medications known to prolong the QT interval while receiving protocol treatment. These medications include selected antiarrhythmics, antihistamines, macrolide antibiotics, and /or tricyclic antidepressants as follows:

Albuterol Alfuzosin Amantadine Amiodarone Amitriptyline Amphetamine Arsenic Trioxide Astemizole Atazanavir Atomoxetine Azithromycin Chloroquine Clomipramine Dolasetron Metaproterenol Moxifloxacin Phenermine Phenylpropanolamine

* Those drugs not specifically listed above but possibly suspected of causing QT prolongation would not necessarily preclude patient registration, but would be discussed with the attending physician prior to initiation of protocol therapy.
* Patients with QTc >450 msec.
* Patients with liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* Patients with acute cholecystitis
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot).
* Patients with abnormal coagulation (INR>1.5) or patients receiving anticoagulants that affect PT (prothrombin time) or APTT ( activated thromboplastin time)
* Patients with WBC <3 K/mcL; PLT < 100 K/mcL
* Patients who have any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the Investigator.
* Patients who have participated in any clinical investigation with an investigational drug (other then pasireotide) within 30 days prior to dosing.
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR or s.c. formulations
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Allen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Allen PJ, Gonen M, Brennan MF, Bucknor AA, Robinson LM, Pappas MM, Carlucci KE, D'Angelica MI, DeMatteo RP, Kingham TP, Fong Y, Jarnagin WR. Pasireotide for postoperative pancreatic fistula. N Engl J Med. 2014 May 22;370(21):2014-22. doi: 10.1056/NEJMoa1313688. PMID 24849084
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- SOM230: This is a randomized, double-blind, placebo controlled phase III trial of SOM230 vs. saline placebo in patients undergoing pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy at MSKCC. Pasireotide (SOM230): Patients will receive subcutaneous injection of SOM230 or placebo (NS, equivalent volume) on the day of operation prior to resection in the pre-surgical center. The initial subcutaneous injection of drug or placebo will be given at least one hour prior but no longer than 8 hours prior to transection of the pancreas. Patients will be continuously monitored in the OR following this dose administration, and both their cardiac and respiratory status will be closely followed. Postoperatively patients will receive study drug or placebo every 12 hours. Subcutaneous injections will continue until postoperative day 7, with the last dose administered in the evening on postoperative day 6, or until a pancreatic complication has been identified.
- Placebo: This is a randomized, double-blind, placebo controlled phase III trial of SOM230 vs. saline placebo in patients undergoing pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy at MSKCC. Patients will receive subcutaneous injection of SOM230 or placebo (NS, equivalent volume) on the day of operation prior to resection in the pre-surgical center. The initial subcutaneous injection of drug or placebo will be given at least one hour prior but no longer than 8 hours prior to transection of the pancreas. Patients will be continuously monitored in the OR following this dose administration, and both their cardiac and respiratory status will be closely followed.
  Postoperatively patients will receive study drug or placebo every 12 hours. Subcutaneous injections will continue until postoperative day 7, with the last dose administered in the evening on postoperative day 6, or until a pancreatic complication has been identified.
Period: Overall Study
Arm/Group | SOM230 | Placebo
Started | 217 | 222
Completed | 152 | 148
Not Completed | 65 | 74
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Not Treated | 4 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Patient not resected | 41 | 52
Not completed — Pt not eligible | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOM230 | Placebo | Total
Number analyzed (Participants) | 217 | 222 | 439
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 104 | 211
  >=65 years | 110 | 118 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 91 | 188
  Male | 120 | 131 | 251
Region of Enrollment [Number; unit: participants]
  United States | 217 | 222 | 439

OUTCOME MEASURES:

1. Primary Outcome: To Compare 60-day ≥Grade 3 Pancreatic Complication Rates (Fistula, Leak, and Abscess) as Defined by the MSKCC Surgical Secondary Events System Between Patients Who Receive Perioperative SOM230 and Saline Placebo.
Time Frame: 60 days
Measure: Number; unit: percentage of participants
Arm/Group | SOM230 | Placebo
Number analyzed (Participants) | 150 | 149
percentage of participants | 9 | 21

ADVERSE EVENTS:
Arm/Group | SOM230 | Placebo
Serious Adverse Events (participants affected / at risk) | 138/217 | 218/222
Other Adverse Events (participants affected / at risk) | 152/217 | 150/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 (N=217) | Placebo (N=222)
Abdominal infection (Infections and infestations) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 11 (11) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 12 (12) | 19 (20)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 1 (2)
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 5 (5) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 89 (90) | 54 (55)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 5 (5) | 4 (4)
Lipase increased (Investigations) | 4 (6) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 8 (8) | 4 (4)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 13 (13) | 20 (20)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 2 (3)
Serum amylase increased (Investigations) | 49 (49) | 36 (36)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 5 (5) | 7 (7)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 6 (6)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 7 (7) | 23 (23)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
INR increase (Investigations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 (N=217) | Placebo (N=222)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 11 (12)
Alanine aminotransferase increased (Investigations) | 47 (181) | 54 (197)
Alkaline phosphatase increased (Investigations) | 22 (107) | 23 (186)
Ascites (Gastrointestinal disorders) | 16 (16) | 26 (29)
Aspartate aminotransferase increased (Investigations) | 47 (98) | 53 (122)
Atrial fibrillation (Cardiac disorders) | 11 (13) | 9 (10)
Blood bilirubin increased (Investigations) | 50 (259) | 56 (243)
Hyperglycemia (Metabolism and nutrition disorders) | 147 (1010) | 130 (746)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (16) | 13 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 66 (325) | 58 (416)
Hypocalcemia (Metabolism and nutrition disorders) | 123 (756) | 125 (849)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (18) | 7 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 123 (271) | 98 (265)
INR increased (Investigations) | 15 (41) | 9 (18)
Lymphocyte count decreased (Investigations) | 56 (160) | 56 (145)
Nausea (Gastrointestinal disorders) | 10 (11) | 13 (13)
Neutrophil count decreased (Investigations) | 29 (44) | 33 (73)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 13 (13) | 22 (22)
Serum amylase increased (Investigations) | 59 (134) | 54 (110)
White blood cell decreased (Investigations) | 24 (114) | 27 (115)
Wound infection (Infections and infestations) | 17 (17) | 26 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes